CLINICAL TRIAL: NCT05636345
Title: An Evaluation of a Public Health Campaign in a High School Setting Targeting Pain Related Knowledge and Beliefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Mrs Jagjit Mankelow, Lecturer in Rehabilitation Science, Teesside University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: teesside university
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Pain, Chronic
Keywords: pain science education; pain knowledge; pain beliefs; experience of education
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: exploratory, single-site, mixed-methods study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): High school students receiving a day of pain science education in multiple formats, lectures, experiential, completing a task which consolidates the information.
  Interventions: Other: pain science education

INTERVENTIONS:
Other: pain science education — A full day of pain science education

SUMMARY:
The beliefs held by students lead to behaviours in response to their pain which can be both helpful or a hindrance to how they manage their pain. The one-day education event aims to educate the cohort on the contemporary scientific understanding of persistent pain. It is hoped this event will result in an improvement in the alignment of beliefs and behaviours to contemporary understanding of persistent pain.

The principal aim is to evaluate the pre-post beliefs about pain following a one-day pain education event.

DETAILED DESCRIPTION:
The students will be asked to complete two questionnaires relating to their understanding of pain. One at the start of the conference and one at the end . The first questionnaire will gather demographic information (age, gender, ethnicity and any history of persistent pain). The following questions will be a series of multiple-choice questions relating to beliefs about persistent pain. The second questionnaire to be completed at the end of the day will be identical to the first, minus the demographic questions. Each questionnaire should take 5-10 minutes to complete. So total involvement in this study will be less than 20 minutes. The questionnaires will be provided in an unmarked brown envelope. The envelope will contain two questionnaires one marked "before" and one marked "after". Participants will be asked to complete the "before" questionnaire at the start of the day and then put it back in their envelope. At the end of the day, they will be asked to complete the "after questionnaire". Participants will keep the envelope with them during the day and at no point will their name or any other identifiable information go on the form. At the end of the day, they will be asked to leave the anonymous envelope in a designated area in the room.

ELIGIBILITY:
Inclusion Criteria: students at one of six schools in Berkshire who had been offered the pain study day.

Aged above 16. Providing consent to participate.

Exclusion Criteria:

Students not providing consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Pain Beliefs Questionnaire (PBQ) | one day
  Helps to identify if participant beliefs are biomedical or biopsychosocial focussed, 12-item (Edwards et al, 1992, Walsh and Radcliffe, 2002). There are 2 scales within the PBQ: the organic beliefs scale has 8 items, with score ranges from 8-48, lower scores indicate less biomedical views and higher scores indicate more biomedical views. The psychological scale within the PBQ has 4 items with a score range of 4-24, a higher score indicates more biopsychosocial beliefs about pain and a lower score indicates less biopsychosocial beliefs.
Concept of Pain Inventory-Adult (COPI-Adult) | one day
  The Concept of Pain Inventory-Adult was designed for assessing knowledge and beliefs about pain science (Pate et al, 2022). It is a 13-item questionnaire. Higher COPI-Adult scores reflect greater alignment with contemporary pain science (Total scores can range from 0-52).
Vignette | one day
  Participants were asked what actions they would take if they had pain with regards to medication, scans, daily activity, exercise and work either based on yes/no answers or four to five multiple choice answers. The percentage of recommendations in keeping with guidelines were measured from 0-100% with lower scores indicating intended behaviours that were not in keeping with guidelines.
Semi-structured interviews | 3 months after the pain education day
  To explore pain beliefs after the education day and experience of the education day.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Anne College, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andias R, Sa-Couto P, Silva AG. Blended-Learning Pain Neuroscience Education and Exercise in High School Students With Chronic Neck Pain: A Randomized Controlled Trial. Phys Ther. 2022 Jun 3;102(6):pzac048. doi: 10.1093/ptj/pzac048. PMID 35485186
- [Background] Neto M, Andias R, Silva AG. Pain Neuroscience Education and Exercise for Neck Pain: A Focus Group Study on Adolescents' Views. Pediatr Phys Ther. 2018 Jul;30(3):196-201. doi: 10.1097/PEP.0000000000000511. PMID 29924066
- [Background] Pate JW, Noblet T, Hush JM, Hancock MJ, Sandells R, Pounder M, Pacey V. Exploring the concept of pain of Australian children with and without pain: qualitative study. BMJ Open. 2019 Oct 28;9(10):e033199. doi: 10.1136/bmjopen-2019-033199. PMID 31662406
- [Background] Pate JW, Simons LE, Rush G, Hancock MJ, Hush JM, Verhagen A, Pacey V. The Concept of Pain Inventory for Adults (COPI-Adult): Assessing Knowledge and Beliefs Regarding Pain Science Education. Clin J Pain. 2021 Oct 12;38(1):32-40. doi: 10.1097/AJP.0000000000000990. PMID 34636751
- [Background] Walsh DA, Radcliffe JC. Pain beliefs and perceived physical disability of patients with chronic low back pain. Pain. 2002 May;97(1-2):23-31. doi: 10.1016/s0304-3959(01)00426-2. PMID 12031776